CLINICAL TRIAL: NCT04477681
Title: Securing Access to Innovative Molecules in Oncology and Hematology for Children, Adolescents and Young Adults in Therapeutic Failure or Relapse and Not Eligible for a Clinical Trial: a Project of the SFCE
Brief Title: Securing Access to Innovative Molecules in Oncology and Hematology for Children, Adolescents and Young Adults
Acronym: SACHA
Status: Recruiting | Type: Observational
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A01317-50; 2019/2848 (Other: CSET number)
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in therapeutic failure or relapse: Any child, adolescent or young adult, treated for a pediatric tumor or leukemia, in therapeutic failure or relapse without standard treatment option, not eligible / refusal of inclusion in a clinical study open on the territory and treated with an innovative drug within the framework of a compassionate use or outside marketing authorization, in one of the centers of the SFCE (Société Française des Cancers de l' Enfant)
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — In particular, the patient's demographic data, medical history, previous and concomitant treatments, data on the treatment of interest (legal framework, compassionate use/ off-label), dosage, start date, etc.), clinical data will be collected. biological (including molecular profiling of the tumor if available) and radiological follow-up, information on adverse effects. The data to be filled in is that of the CERFA pharmacovigilance form of the ANSM, but additional fields can be created if necessary.

SUMMARY:
It involves collecting safety and efficacy data, under the actual conditions of use of medicines in children and adolescents, using a validated tool (Ennov EDC) and relying on the network of Interregional pediatric oncology appeal organizations (RIOs) identified by INCa since 2010 and responsible for the organization of Pluridisciplinary Pediatric Interregional (RCPPI) and National Consultative Meetings which discuss each case of relapse in order to define the best therapeutic options.

DETAILED DESCRIPTION:
The objective is to aim for completeness throughout the national territory. This is why this project will be carried out in close collaboration with the RIOs and RCPPI and that of the 31 centers of the SFCE which bring together more than 400 doctors pediatric oncologists and hematologists on the French territory

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 25 years old at the time of inclusion in the study
* Patient with a pediatric tumor or leukemia in therapeutic failure or relapse without standard therapeutic options. Exceptionally, patients on the first line of treatment without standard therapeutic options may also be included (eg g: inoperable plexiform neurofibroma and MEK inhibitors, childhood fibrosarcoma and NTRK inhibitors).
* Patient not eligible for an early phase clinical trial open to inclusion on French territory or refusal of inclusion
* Patient treated with a new drug discussed at a RCPPI as part of a compassionate use issued by the ANSM or an off-label prescription of a drug of interest already authorized in adults.
* Patients treated in one of the SFCE centers authorized to prescribe chemotherapy
* Patient who did not object to participate after being informed of the study. The patient must be able and willing to cooperate in the study.

Exclusion Criteria:

* Patient included in an early phase clinical trial open to inclusions on French territory.
* Oral refusal to participate by the patient or their legal representatives, in reading the information note specific to the study
* Patient under guardianship or curatorship, deprived of liberty or in the impossibility of expressing opposition to participating in the study

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any child, adolescent or young adult, treated for a pediatric tumor or leukemia, in therapeutic failure or relapse without standard treatment option, not eligible / refusal of inclusion in a clinical study open on the territory and treated with an innovative drug within the framework of compassionate use or outside marketing authorization, in one of the centers of the SFCE (Société Française des Cancers de l' Enfant).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Collect access data | up to 1 year
  Collect access data of children, adolescents and young adults in therapeutic failures and not eligible for a clinical trial with innovative molecules, whether they are targeted therapies, immunotherapies or chemotherapies

CONTACTS AND LOCATIONS:
Locations (31):
- France (31):
  - Gustave Roussy, Villejuif, Val De Marne
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU CAEN, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - Centre Oscar Lambret, Lille
  - CHU Lille, Lille
  - CHU Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - CHU Lyon, Lyon
  - Hôpital de La Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Hôpital Armand Trousseau, Paris
  - Hôpital Robert-Debré, Paris
  - Institut Curie, Paris
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU La Réunion, Saint-Denis
  - CHU Saint-Etienne, Saint-Etienne
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berlanga P, Ndounga-Diakou LA, Aerts I, Corradini N, Ducassou S, Strullu M, de Carli E, Andre N, Entz-Werle N, Raimbault S, Roumy M, Renouard M, Gueguen G, Plantaz D, Reguerre Y, Cleirec M, Petit A, Puiseux C, Andry L, Klein S, Bodet D, Kanold J, Briandet C, Halfon-Domenech C, Nelken B, Piguet C, Saumet L, Chastagner P, Benadiba J, Millot F, Pluchart C, Schneider P, Thouvenin S, Gambart M, Serre J, Abbou S, Leruste A, Cayzac H, Gandemer V, Laghouati S, Vassal G. Measuring Safety and Outcomes for the Use of Compassionate and Off-Label Therapies for Children, Adolescents, and Young Adults With Cancer in the SACHA-France Study. JAMA Netw Open. 2023 Jul 3;6(7):e2321568. doi: 10.1001/jamanetworkopen.2023.21568. PMID 37399010
- [Derived] Pasqualini C, Proust S, Schleiermacher G, Gambart M, Jannier S, Petit A, Dupraz C, Thebaud E, Reguerre Y, Ndounga-Diakou LA, Laghouat S, Defachelles AS, Berlanga P. Chemo-Immunotherapy Rescue for High-Risk Neuroblastoma Patients With Progressive Disease Before High-Dose Chemotherapy: Real-World Data From the SACHA-France Study. Pediatr Blood Cancer. 2025 Dec;72(12):e32080. doi: 10.1002/pbc.32080. Epub 2025 Oct 3. PMID 41044876
- See also: Institutional website (Gustave Roussy) — https://www.gustaveroussy.fr/fr/sacha